CLINICAL TRIAL: NCT06993233
Title: A Phase 2a Double Blind, Randomized, Parallel Arm, Placebo-controlled Trial to Investigate the Effects of Two Dose Levels of CIT-013 on Disease Activity in Patients With Hidradenitis Suppurativa
Brief Title: A Study With CIT-013 in HS Patients
Acronym: Citylights
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Citryll BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CITRYLL003
Record Dates: First submitted 2025-05-19; First posted 2025-05-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CIT-013 high dose (Experimental): 6 SC injections with CIT-013 high dose
  Interventions: Drug: CIT-013 high dose
- CIT-013 medium dose (Experimental): 6 SC injections with CIT-013 medium dose
  Interventions: Drug: CIT-013 medium dose
- Placebo (Placebo Comparator): 6 SC injections with placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CIT-013 high dose — subcutaneous injection
  Arms: CIT-013 high dose
Drug: CIT-013 medium dose — subcutaneous injection
  Arms: CIT-013 medium dose
Drug: Placebo — subcutaneous injection
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if CIT-013 works to treat Hidradenitis Suppurativa in adults. It will also learn about the safety of CIT-013. The main questions it aims to answer are:

Does CIT-013 lower the disease activity of HS patients? What medical problems do participants have when receiving CIT-013? Researchers will compare CIT-013 to a placebo (a look-alike substance that contains no drug) to see if CIT-013 works to treat the symptoms of HS.

Participants will:

Take receive 50 or 100 mg CIT-013 or placebo every other week for 12 weeks Visit the clinic once every 2 weeks for checkups and tests Keep monitor their symptoms during this period

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with HS of more than 6 months duration,
* 18 years of age at screening visit,
* Hidradenitis suppurativa lesions present in ≥ 2 distinct anatomic areas, one of which is Hurley Stage II or III (according to Hurley classification system),
* A total abscess and inflammatory nodule (AN) count of ≥ 5 at screening and Day 1 prior to enrollment/randomization,
* Participant must have had an inadequate response to oral antibiotics OR exhibited recurrence after discontinuation to, OR demonstrated intolerance to, OR have a contraindication to oral antibiotics for treatment of their HS,
* Total draining tunnel count less than 20

Exclusion Criteria:

- Participants for whom an approved therapy with demonstrated clinical benefit is indicated, available and expected to be tolerated, OR choose to proceed with standard of care treatment options over the IP (after being appropriately informed of the treatment options, risks, and benefits).

Any current and/or recurrent clinically significant skin condition in the treatment area other than HS,

* Prior treatment with a recombinant therapeutic protein during the 6 weeks before baseline
* Prior treatment with any of the following medications before baseline:

  1. Any other systemic therapy for HS (28 days before baseline)
  2. Any IV anti-infective therapy (14 days before baseline)
* History of malignancy with exception of non-melanoma skin cancer that has been excised and cured,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with HiSCR75 on CIT 013 versus placebo | week 12

SECONDARY OUTCOMES:
Incidence of TEAEs as assessed by CTCAE | week 12
Maximum Plasma Concentration of CIT-013 before doses | 4, 6, 10 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Kraan, Study Director — Citryll BV
Locations (24):
- Canada (5):
  - CA-01, Barrie
  - CA-05, Calgary
  - CA-02, London
  - CA-04, Newmarket
  - CA-03, Winnipeg
- Germany (6):
  - DE-06, Bad Bentheim
  - DE-01, Bochum
  - DE-04, Dresden
  - DE-02, Frankfurt
  - DE-08, Kiel
  - DE-03, Oldenburg
- Erasmus UMC, Rotterdam, Netherlands
- Poland (4):
  - PL-03, Katowice
  - PL-02, Lodz
  - PL-01, Rzeszów
  - PL-05, Wroclaw
- Spain (5):
  - ES-05, Barcelona
  - ES-04, Madrid
  - ES-02, Santiago de Compostela
  - ES-03, Seville
  - ES-01, Valencia
- United Kingdom (3):
  - GB-02, Cardiff
  - GB-05, Chester
  - GB-04, London